CLINICAL TRIAL: NCT04788394
Title: Renal Involvement in Hospitalized Children With COVID-19
Acronym: RIHCC
Status: Completed | Type: Observational
Sponsor: Hamad Medical Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: MRC01-21-089
Record Dates: First submitted 2021-03-07; First posted 2021-03-09 (Actual); Last update posted 2023-07-25 (Actual); Status verified 2021-03

CONDITIONS: Acute Kidney Injury; Covid19; Renal Dysfunction; Coronavirus Infection; AKI; Pediatric Kidney Disease; Renal Insufficiency
MeSH Terms: conditions — Acute Kidney Injury; COVID-19; Renal Insufficiency; Coronavirus Infections

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: data review — In this retrospective study investigators will include all children and adolescents (≤ 18 years old) with pre-existing CKD and laboratory confirmed SARS-CoV-2 infection who were treated at Hamad General Hospital, in Doha, Qatar during this pandemic using the electronic medical records since 1st March 2020 till January 20th, 2022. Indications for testing patients for SARS CoV-2 infection included:
  * Clinical features suggestive of COVID-19 (fever, cough, dyspnea, rhinorrhea, sore throat, diarrhea, myalgia, anosmia, or ageusia).
  * Close contact (within 6-ft of an infected person for 15 min or longer) within an individual diagnosed with SARS-CoV-2 infection [40].
  * Admission for management of the underlying disease. le against the age-specific upper limit of reference interval (ULRI) values according to Hamad Hospital guidelines. Acute kidney injury will be defined as a serum creatinine 1.5 times greater than the ULRI.
  to determine:
Other: data comparing — In this retrospective study investigators will include all children and adolescents (≤ 18 years old) with pre-existing CKD and laboratory-confirmed SARS-CoV-2 infection who were treated at Hamad General Hospital, in Doha, Qatar during this pandemic using the electronic medical records since 1st March 2020 till January 20th, 2022. Indications for testing patients for SARS CoV-2 infection included:
  * Clinical features suggestive of COVID-19 (fever, cough, dyspnea, rhinorrhea, sore throat, diarrhea, myalgia, anosmia, or ageusia).
  * Close contact (within 6-ft of an infected person for 15 min or longer) within an individual diagnosed with SARS-CoV-2 infection [40].
  * Admission for management of the underlying disease. le against the age-specific upper limit of reference interval (ULRI) values according to Hamad Hospital guidelines. Acute kidney injury will be defined as a serum creatinine 1.5 times greater than the ULRI.
  to determine:

SUMMARY:
Covid-19 is an important human and animal pathogen, it mostly causes respiratory and gastrointestinal symptoms. Clinical features range from a common cold to severe diseases such as severe acute respiratory distress syndrome, bronchitis, pneumonia, multi-organ failure, and even death. It seems to be less commonly affecting children and to cause fewer symptoms and less severe disease in this age group compared with adults. Clinicians have observed many extrapulmonary manifestations of COVID-19, as hematologic, cardiovascular, renal, gastrointestinal and hepatobiliary, endocrinologic, neurologic, ophthalmologic, and dermatologic systems can all be affected. This retrospective study that will be conducted at Hamad General Hospital in Qatar, aims to determine the renal involvement in all pediatric patients who were hospitalized with COVID-19 from March 1, 2020, to January 1, 2021.

DETAILED DESCRIPTION:
COVID-19 usually causes respiratory and gastrointestinal symptoms, Clinical features range from a common cold to severe diseases such as bronchitis, pneumonia, severe acute respiratory distress syndrome, multi-organ failure, and even death. SARS-CoV, MERS-CoV, and SARS-CoV-2 seem to less commonly affect children and to cause fewer symptoms and less severe disease in this age group compared with adults and are associated with much lower case-fatality rates. Coronaviruses are a large family of enveloped, single-stranded, zoonotic RNA viruses. Clinicians have observed many extrapulmonary manifestations of COVID-19, as hematologic, cardiovascular, renal, and gastrointestinal and hepatobiliary, endocrinologic, neurologic, ophthalmologic, and dermatologic systems can all be affected.

Acute kidney injury (AKI) is a frequent complication of COVID-19 and is associated with mortality. In adults, the incidence of AKI in hospitalized patients with COVID-19 ranged from 0.5% to 29% and occurred within a median of 7-14 days after admission. Studies from the USA have reported much higher rates of AKI. In a study of nearly 5,500 patients admitted with COVID-19 in a New York City hospital system, AKI occurred in 37%, with 14% of the patients requiring dialysis. AKI occurred at much higher rates in critically ill patients admitted to New York City hospitals, ranging from 78% to 90%. Of 257 adult patients admitted to ICUs in a study from New York City, 31% received renal replacement therapy (RRT). Furthermore, hematuria has been reported in nearly half of patients with COVID-19, and proteinuria has been reported in up to 87% of critically ill patients with COVID-19 (11). Hyperkalemia and acidosis are common electrolyte abnormalities seen in patients with COVID-19, even among patients without AKI. COVID-19 is also increasingly reported among patients with end-stage renal disease and kidney transplant recipients, with higher mortality rates than those seen in the general population.

Children and adolescents with COVID-19 fare considerably better than adults, with mortality rates in pediatric patients (age <18 years) of less than 1% reported in early studies . The most common clinical features in children described in the literature are fever, dry cough, and pneumonia . However, multisystem involvement is increasingly being recognized, including the development of hyperinflammatory shock.

In other studies, acute kidney injury has been reported in adult patients with COVID-19, with a high prevalence across inpatient admissions (≤7%) and admissions to adult intensive care units (ICUs; ≤23%), as first reported in Wuhan, China . In adult patients with COVID-19, acute kidney injury is related to increased mortality risk, even after adjustment for age, sex, and comorbidities. In addition, a large proportion of adults have proteinuria (44%) and hematuria (27%) at presentation, despite an elevated serum creatinine prevalence of only 16% .

In children, there is scanty data compared to adults, Douglas et al studied 52 pediatric patients (ages 0-16 years) admitted to Great Ormond Street Hospital for Children NHS Foundation Trust (London, UK) since March 25, 2020, with confirmed severe acute respiratory syndrome coronavirus infection, and diagnosed by either a positive PCR result or seropositivity. Of the 52 inpatients, 24 (46%) had a serum creatinine greater than the upper limit of reference interval (ULRI), 22 [42%] had proteinuria, and hematuria was found in 40 [77%] patients. Qui and colleagues (18) did not find any renal dysfunction in 36 hospitalized pediatric patients (ages 0-16 years) with COVID-19 in China. Renal dysfunction defined by a serum creatinine greater than 110 μmol/L or serum urea greater than 7 mmol/L.

This retrospective, exploratory, descriptive study aims to determine the renal involvement in all pediatric patients who were hospitalized with COVID-19 in Qatar.

ELIGIBILITY:
Inclusion Criteria:

All pediatric patients with COVID-19 were admitted to Hamad Hospital from (0 to 14) years, using the electronic medical records (Cerner), over that time period (from March 1, to January 1, 2021), with one of the following:

* Proteinuria: (≥1+) on dipstick analysis.
* Hematuria: ≥ 5 RBC/HPF.
* Sterile Pyuria: ≥ 5 WBC/HPF or ≥10 WBC/mm3 with negative urine culture (44).
* Hypernatremia :> 145meq/l.
* Hyponatremia: < 135 meq/l.
* Hypokalemia :< 3.5meq/l.
* Metabolic acidosis (ph <7.35).
* Elevated serum creatinine :> upper limit of reference interval (ULRI) values.
* Elevated serum urea: > 7 mmol/l.
* Urine specific gravity (SG) <1.003.

Exclusion Criteria:

* Patient with previous chronic kidney diseases.

Ages: 1 Day to 14 Years | Sex: All
Age Groups: Child
Study Population: This retrospective review of electronic medical records from the pediatric division, Hamad General hospital in Doha, Qatar, will include all hospitalized children (0-14 years) who were diagnosed with COVID-19 between March 1, 2020, to January 1, 2021. Data collection will be done by co-investigators for all patients.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
determine the prevalence of renal dysfunction in hospitalized children with COVID19 in Qatar. | 1 year
  explore and describe the rate of renal symptoms and signs, and severity in pediatric patients admitted to the hospital with COVID 19 in Qatar . The relation between severity of disease and age , weight , gender ,and nationality of participants .

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud Alhandi Omar Helal, Principal Investigator — Hamad Medical Corporation; Mahmoud Helal, Principal Investigator — Hamad Medical Corporation
Locations (1):
- Hamad General corporation, Doha, Qatar